CLINICAL TRIAL: NCT00471562
Title: Phase I Clinical Trial of Angiotensin 1-7 for Advanced Solid Tumors
Brief Title: Angiotensin-(1-7) in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000543744; CCCWFU-99206; CCCWFU-99206/Ang 1-7; CCCWFU-IRB00001136; NCT01581268 (obsolete NCT alias)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — angiotensin I (1-7)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: therapeutic angiotensin-(1-7) — sequentially increasing doses 50-1000 mcg/kg

SUMMARY:
RATIONALE: Angiotensin-(1-7) may stop the growth of solid tumors by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of angiotensin-(1-7) in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of therapeutic angiotensin-(1-7) in patients with metastatic or unresectable solid tumors.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine tumor response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive therapeutic angiotensin-(1-7) subcutaneously on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of therapeutic angiotensin-(1-7) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first 3 weeks of study therapy. At least 6 patients are treated at the MTD.

Blood samples are collected from patients after the first and fifth doses of the study drug for pharmacokinetic correlative studies.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor meeting 1 of the following criteria:

  * Metastatic disease
  * Unresectable disease
* Standard curative or palliative measures do not exist or are no longer effective
* Measurable or nonmeasurable disease

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
  * Nonmeasurable disease, defined as all other lesions, including small lesions (i.e., ≥ 1 unidimensionally measurable lesion < 20 mm by conventional techniques or < 10 mm by spiral CT scan) and truly nonmeasurable lesions, including any of the following:

    * Bone lesions
    * Ascites
    * Pleural or pericardial effusion
    * Lymphangitis cutis or pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No lung cancer with recent hemoptysis
* No brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 4 weeks
* No evidence of bleeding diathesis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance > 30 mL/min
* Bilirubin < 2 mg/dL
* AST and ALT < 3 times upper limit of normal
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Uncontrolled hypertension or hypotension
* No psychiatric illness or social situation that would preclude informed consent or study compliance

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior major surgery
* At least 4 weeks since prior radiotherapy or chemotherapy (6 weeks for melphalan, nitrosoureas, or mitomycin C)
* No concurrent therapeutic anticoagulation
* No other concurrent investigational agents
* No concurrent angiotensin-converting enzyme inhibitors or angiotensin II receptor blockers
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 21 days
Toxicity | 105 days

SECONDARY OUTCOMES:
Response rate (complete or partial response) as measured by RECIST criteria | 105 days

CONTACTS AND LOCATIONS:
Overall Officials: W. Jeffrey Petty, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Petty WJ, Miller AA, McCoy TP, Gallagher PE, Tallant EA, Torti FM. Phase I and pharmacokinetic study of angiotensin-(1-7), an endogenous antiangiogenic hormone. Clin Cancer Res. 2009 Dec 1;15(23):7398-404. doi: 10.1158/1078-0432.CCR-09-1957. Epub 2009 Nov 17. PMID 19920106